CLINICAL TRIAL: NCT01929551
Title: Comparison of the Glycemic Index of a Drink Made of Natural Concentrated Mango Puree With Natural Concentrated Pear Juice With That of Other Five Products Based on Mango and Pear in Different Solid Products and Drinks
Brief Title: Glycemic Index of Mango and Pear in Different Solid Products and Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Leticia Elizondo-Montemayor, M.D., Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: IGPMJP2013-CINCO
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-09

CONDITIONS: Glucose Intolerance
Keywords: glycemic index
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Mango puree and pear juice beverage (Other): Participants will drink 450 milliliters of the juice at time 0.
  Interventions: Other: Mango puree and pear juice beverage
- Commercial mango juice (Other): Participants will drink 450 milliliters of the juice at time 0.
  Interventions: Other: Commercial mango juice
- Fresh natural mango (Other): Participants will eat 400 to 500 grams of frozen mango pulp, along with 250 milliliters of water at time 0.
  Interventions: Other: Fresh natural mango
- Frozen natural mango (Other): Participants will eat 400 to 500 grams of frozen mango pulp, along with 250 milliliters of water at time 0.
  Interventions: Other: Frozen natural mango
- Processed natural mango pulp (Other): Participants will eat 400 to 500 grams of frozen mango pulp, along with 250 milliliters of water at time 0.
  Interventions: Other: Processed natural mango pulp
- Mix of natural mango and pear (Other): Participants will eat 400 to 500 grams of a mixture of fresh natural fruit containing mango (73%) and pear (27%), along with 250 milliliters of water at time 0.
  Interventions: Other: Mix of natural mango and pear
- 50 grams glucose load (Other): Participants will drink 250 milliliters of the standard glucose load at time 0.
  Interventions: Other: 50 grams glucose load

INTERVENTIONS:
Other: Mango puree and pear juice beverage — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index of MPPJB.
  Arms: Mango puree and pear juice beverage
Other: Commercial mango juice — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index of commercial mango juice
  Arms: Commercial mango juice
Other: Fresh natural mango — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index of fresh natural mango
  Arms: Fresh natural mango
Other: Frozen natural mango — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index of frozen natural mango
  Arms: Frozen natural mango
Other: Processed natural mango pulp — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index of PNMP.
  Arms: Processed natural mango pulp
Other: Mix of natural mango and pear — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index for mix of NMP.
  Arms: Mix of natural mango and pear
Other: 50 grams glucose load — Capillary glucose will be taken every 15 minutes for two hours (starting at time 0) to calculate the area under the curve which is the glycemic index, for each of the products.
  Other Names: Determination of glycemic index for 50 grams glucose load
  Arms: 50 grams glucose load

SUMMARY:
The purpose of this study is to compare the glycemic index of a beverage made of natural concentrated mango puree with natural concentrated pear juice with other five different products based on natural mango and pear ingredients in the form of fruit or juice against a control of 50-gram glucose load.

DETAILED DESCRIPTION:
The participants will be recruited with an open invitation to participate, those who voluntarily accept, sign an informed consent, and meet the all inclusion criteria and none of the exclusion criteria will participate.

Each participant will receive a different product (of the seven products available) each day of the test (8 days in total), making sure everyone receives each one of the products. All products will be distributed in a randomized fashion for each of the participants. The 50-gram glucose load (gold standard) will be the reference or control, and will be taken twice by each subject in the test.

Each one of the products given will contain 50 grams of carbohydrate. The time given to consume the products will be 10 minutes total.

There will be a "wash out" period of three days in between each product.

The participants will eat the product and capillary glucose will be taken with a glucometer (Accu-Chek Performa System © 2009 Roche Diagnostics. Roche Products, México) at times: 0, 15, 30, 45, 60, 75, 90, 150 and 120 minutes. The glucometer will be calibrated with a standard glucose solution every day previous to the test. The results will be used to calculate the glycemic index. At the end of the 120 minutes, the participants will receive a questionnaire of digestive symptoms presented during the test.

The glycemic index will be calculated by the area under the curve for each product divided by the area under the curve for the 50-gram glucose load, multiplied by 100. The area under the curve used to calculate the glycemic index is the area that surpasses the basal line, excluding the area under the basal line according to the Food and Agriculture Organization (FAO) in 1998 (Brouns et al 2005).

All information collected will be emptied into a pre-designed database.

The differences between the different products ingested will be analyzed with the statistical test of analysis of variance (ANOVA) with a pre-test of homogeneity of variance Brown-Foryhte. In case of failure to find homogeneity in the variances the nonparametric ANOVA, the Kruskal-Wallis test, will be used. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.

After ANOVA, Tuckey Multiple Comparisons test will be used to evaluate the pairwise relationship for each product.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Ages 18 to 50 years
* Body mass index between 18.5 and 27.4 kilograms divided by squared meters
* Waist circumference ≤ 102 centimeters for men and ≤88 centimeters for women
* Fasting capillary glucose ≤100 milligrams per deciliter

The night before the study:

* 10 hours fasting
* Light dinner of their choice and repeat it every time before the study
* No alcohol, coffee or tea drinks the previous night
* No vigorous exercise the day before the test nor the morning of the test

Exclusion Criteria:

* Consumption of any of the following: oral hypoglycemic drugs, oral or parenteral glucocorticoid drugs, thyroid hormones, stimulant of intestinal motility or other drugs that may interfere with the intestinal absorption during the test
* Acute or chronic gastrointestinal infections
* Breast feeding or pregnant women
* Intestinal surgeries in the last 6 months
* Allergies to any of the products we will be using
* Subjects with gastrointestinal or metabolic diseases
* Subjects with first grade family history of diabetes mellitus
* Subjects with glucose intolerance, insulin resistance or diabetes mellitus
* Subjects who dislike any of the products we will be using
* Subjects with an acute (previous 24 hours) digestive crisis including: gastritis, diarrhea, and vomit, among others
* Subjects with a history of mal-absorption

Suspension:

* Subjects that do not arrive at the test-day
* Fasting glucose ≥ 100 milligrams per deciliter the day of the test
* Subjects who develop gastrointestinal disease during the study time frame

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Glycemic index of mango puree with natural pear juice beverage | 8 days
  Glycemic index will be calculated for 450 milliliters of this juice. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.

SECONDARY OUTCOMES:
Glycemic index of a commercial mango juice | 8 days
  Glycemic index will be calculated for 450 milliliters of this juice. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.
Glycemic index of natural fresh mango | 8 days
  Glycemic index will be calculated for 400 to 500 grams of mango along with 250 milliliters of water. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.
Glycemic index of natural frozen mango pulp | 8 days
  Glycemic index will be calculated for 400 to 500 grams of mango along with 250 milliliters of water. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.
Glycemic index of processed natural mango pulp | 8 days
  Glycemic index will be calculated for 400 to 500 grams of mango along with 250 milliliters of water. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.
glycemic index of a mixture of fresh mango 73 percent and fresh pear 27 percent | 8 days
  Glycemic index will be calculated for 400 to 500 grams of mango along with 250 milliliters of water. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.
glycemic index of a 50 gram glucose load | 8 days
  Glycemic index will be calculated for a standard 50-gram glucose load. This will be done twice by every participant. The results will be expressed as mean ± standard deviation for each with a significance level of 0.05 for all the statistical tests.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Elizondo-Montemayor, MD, Principal Investigator — Clinical Nutrition and Obesity Research Center. TEC Salud, School of Medicine and Health Sciences. Instituto Tecnologico y de Estudios Superiores de Monterrey
Locations (1):
- Clinical Nutrition and Obesity Research Center. School of Medicine and Health Sciences, TEC Salud, Tecnológico de Monterrey, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Brand JC, Holt S, Saveny and Hanksy J. Plasma glucose correlates inversely with satiety and CCK. Proc Nutr Soc Aust 1990; 15: 209 (abstr).
- [Background] Brock DW, Davis CK, Irving BA, Rodriguez J, Barrett EJ, Weltman A, Taylor AG, Gaesser GA. A high-carbohydrate, high-fiber meal improves endothelial function in adults with the metabolic syndrome. Diabetes Care. 2006 Oct;29(10):2313-5. doi: 10.2337/dc06-0917. No abstract available. PMID 17003313
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901
- [Background] Carlson JJ, Eisenmann JC, Norman GJ, Ortiz KA, Young PC. Dietary fiber and nutrient density are inversely associated with the metabolic syndrome in US adolescents. J Am Diet Assoc. 2011 Nov;111(11):1688-95. doi: 10.1016/j.jada.2011.08.008. PMID 22027051
- [Background] Carlson JJ, Monti V. The role of inclusive dietary patterns for achieving secondary prevention cardiovascular nutrition guidelines and optimal cardiovascular health. J Cardiopulm Rehabil. 2003 Sep-Oct;23(5):322-33. doi: 10.1097/00008483-200309000-00001. No abstract available. PMID 14512776
- [Background] Carlson JJ, Winkleby M, Gardner C, Ahn D. Plant-based food intake and cardiovascular disease (CVD) risk factor status in a national sample of ethnically diverse women (NHANES III) FASEB J. 2003a;17:A372.
- [Background] Delzenne NM, Cani PD. A place for dietary fibre in the management of the metabolic syndrome. Curr Opin Clin Nutr Metab Care. 2005 Nov;8(6):636-40. doi: 10.1097/01.mco.0000171124.06408.71. PMID 16205465
- [Background] Dubnov-Raz G, Berry EM. The dietary treatment of obesity. Endocrinol Metab Clin North Am. 2008 Dec;37(4):873-86. doi: 10.1016/j.ecl.2008.08.002. PMID 19026937
- [Background] Ellison JM, Stegmann JM, Colner SL, Michael RH, Sharma MK, Ervin KR, Horwitz DL. Rapid changes in postprandial blood glucose produce concentration differences at finger, forearm, and thigh sampling sites. Diabetes Care. 2002 Jun;25(6):961-4. doi: 10.2337/diacare.25.6.961. PMID 12032099
- [Background] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Background] Granfeldt Y, Hagander B, Bjorck I. Metabolic responses to starch in oat and wheat products. On the importance of food structure, incomplete gelatinization or presence of viscous dietary fibre. Eur J Clin Nutr. 1995 Mar;49(3):189-99. PMID 7774535
- [Background] Halton TL, Willett WC, Liu S, Manson JE, Albert CM, Rexrode K, Hu FB. Low-carbohydrate-diet score and the risk of coronary heart disease in women. N Engl J Med. 2006 Nov 9;355(19):1991-2002. doi: 10.1056/NEJMoa055317. PMID 17093250
- [Background] Hatonen KA, Simila ME, Virtamo JR, Eriksson JG, Hannila ML, Sinkko HK, Sundvall JE, Mykkanen HM, Valsta LM. Methodologic considerations in the measurement of glycemic index: glycemic response to rye bread, oatmeal porridge, and mashed potato. Am J Clin Nutr. 2006 Nov;84(5):1055-61. doi: 10.1093/ajcn/84.5.1055. PMID 17093157
- [Background] Hu FB. Diet and cardiovascular disease prevention the need for a paradigm shift. J Am Coll Cardiol. 2007 Jul 3;50(1):22-4. doi: 10.1016/j.jacc.2007.04.027. Epub 2007 Jun 18. No abstract available. PMID 17601540
- [Background] Hu FB. Plant-based foods and prevention of cardiovascular disease: an overview. Am J Clin Nutr. 2003 Sep;78(3 Suppl):544S-551S. doi: 10.1093/ajcn/78.3.544S. PMID 12936948
- [Background] Jenkins DJ, Wolever TM, Ocana AM, Vuksan V, Cunnane SC, Jenkins M, Wong GS, Singer W, Bloom SR, Blendis LM, et al. Metabolic effects of reducing rate of glucose ingestion by single bolus versus continuous sipping. Diabetes. 1990 Jul;39(7):775-81. doi: 10.2337/diab.39.7.775. PMID 2191884
- [Background] Katcher HI, Legro RS, Kunselman AR, Gillies PJ, Demers LM, Bagshaw DM, Kris-Etherton PM. The effects of a whole grain-enriched hypocaloric diet on cardiovascular disease risk factors in men and women with metabolic syndrome. Am J Clin Nutr. 2008 Jan;87(1):79-90. doi: 10.1093/ajcn/87.1.79. PMID 18175740
- [Background] Kromhout D, Menotti A, Kesteloot H, Sans S. Prevention of coronary heart disease by diet and lifestyle: evidence from prospective cross-cultural, cohort, and intervention studies. Circulation. 2002 Feb 19;105(7):893-8. doi: 10.1161/hc0702.103728. No abstract available. PMID 11854133
- [Background] McCaffrey TA, Rennie KL, Kerr MA, Wallace JM, Hannon-Fletcher MP, Coward WA, Jebb SA, Livingstone MB. Energy density of the diet and change in body fatness from childhood to adolescence; is there a relation? Am J Clin Nutr. 2008 May;87(5):1230-7. doi: 10.1093/ajcn/87.5.1230. PMID 18469244
- [Background] Newby PK, Muller D, Hallfrisch J, Qiao N, Andres R, Tucker KL. Dietary patterns and changes in body mass index and waist circumference in adults. Am J Clin Nutr. 2003 Jun;77(6):1417-25. doi: 10.1093/ajcn/77.6.1417. PMID 12791618
- [Background] Olaiz-Fernández, G., Rivera-Dommarco, J., Shamah-Levy, T., Rojas, R., Villalpando-Hernández, S., Hernández-Avila, M. & Sepúlveda, J. (2006) Encuesta Nacional de Salud y Nutrición. Cuernavaca, México: Instituto Nacional de Salud Pública. Available at: http://www.insp.mx/images/stories/ENSANUT/Docs/Ensanut2006.pdf (Accessed on June 2011)
- [Background] Pan Y, Pratt CA. Metabolic syndrome and its association with diet and physical activity in US adolescents. J Am Diet Assoc. 2008 Feb;108(2):276-86; discussion 286. doi: 10.1016/j.jada.2007.10.049. PMID 18237576
- [Background] Rakel: Integrative Medicine, 2nd ed. Saunders, Elsevier, 2007.
- [Background] Roberts CK, Liu S. Carbohydrate intake and obesity: an association that needs "refining". J Am Diet Assoc. 2009 Jul;109(7):1163-4. doi: 10.1016/j.jada.2009.04.016. No abstract available. PMID 19559131
- [Background] Siri-Tarino PW, Sun Q, Hu FB, Krauss RM. Saturated fat, carbohydrate, and cardiovascular disease. Am J Clin Nutr. 2010 Mar;91(3):502-9. doi: 10.3945/ajcn.2008.26285. Epub 2010 Jan 20. PMID 20089734
- [Background] Steffen LM, Jacobs DR Jr, Murtaugh MA, Moran A, Steinberger J, Hong CP, Sinaiko AR. Whole grain intake is associated with lower body mass and greater insulin sensitivity among adolescents. Am J Epidemiol. 2003 Aug 1;158(3):243-50. doi: 10.1093/aje/kwg146. PMID 12882946
- [Background] Steffen LM, Jacobs DR Jr, Stevens J, Shahar E, Carithers T, Folsom AR. Associations of whole-grain, refined-grain, and fruit and vegetable consumption with risks of all-cause mortality and incident coronary artery disease and ischemic stroke: the Atherosclerosis Risk in Communities (ARIC) Study. Am J Clin Nutr. 2003 Sep;78(3):383-90. doi: 10.1093/ajcn/78.3.383. PMID 12936919
- [Background] Wang Y, Beydoun MA. The obesity epidemic in the United States--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: a systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28. doi: 10.1093/epirev/mxm007. Epub 2007 May 17. PMID 17510091
- [Background] Weickert MO, Pfeiffer AF. Metabolic effects of dietary fiber consumption and prevention of diabetes. J Nutr. 2008 Mar;138(3):439-42. doi: 10.1093/jn/138.3.439. PMID 18287346
- [Background] Wolever TM, Jenkins DJ, Jenkins AL, Josse RG. The glycemic index: methodology and clinical implications. Am J Clin Nutr. 1991 Nov;54(5):846-54. doi: 10.1093/ajcn/54.5.846. PMID 1951155
- [Background] Wolever TM, Mehling C. High-carbohydrate-low-glycaemic index dietary advice improves glucose disposition index in subjects with impaired glucose tolerance. Br J Nutr. 2002 May;87(5):477-87. doi: 10.1079/BJNBJN2002568. PMID 12010586
- [Background] Zehner, L and Zehner W. Mixtures of fructose, sucrose and lactose as a low-calorie bulk sweetener with reduced glycemic index. United States Patent 7560443, 2003.